CLINICAL TRIAL: NCT03099005
Title: Effect of Cannabis Administration and Endocannabinoids on HIV Neuropathic Pain Primary Study - Phase 2
Brief Title: Effect of Cannabis and Endocannabinoids on HIV Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brook Henry, Assistant Research Scientist, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170510
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Cannabis; HIV Neuropathy; Pain Syndrome
Keywords: neuropathic pain; human immunovirus; vaporized cannabis
MeSH Terms: conditions — Marijuana Abuse; Somatoform Disorders; Neuralgia | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Acutely administered CBD/THC will reduce HIV-neuropathic pain in a stair-step manner; the highest CBD dose will provide the greatest pain reduction (high CBD > medium CBD > low CBD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will receive vaporized cannabis using Volcano vaporizers (Storz and Bickel) with either 3.74% THC + 0.49% CBD, 3.49% THC + 4.17% CBD, or 3.11% THC + 15.76% CBD at each of three visits. Allocation assignment of visits will be assigned using a Web-based random number- generating program, "Research Randomizer" (http:// www.randomizer.org/). The allocation schedule will be kept in the pharmacy and concealed from other study personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low CBD session (Active Comparator): In the morning, participants will inhale 8 puffs of vaporized cannabis containing 1.9% THC + 0.01% CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Interventions: Drug: Cannabis
- Medium CBD session (Active Comparator): In the morning, participants will inhale 8 puffs of vaporized cannabis 4 puffs will contain 1.9% THC + 0.01% CBD and 4 puffs will contain 1.4% THC + 5.1% CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Interventions: Drug: Cannabis
- High CBD session (Active Comparator): In the morning, participants will inhale 8 puffs of vaporized cannabis containing 1.4% THC + 5.1% CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — vaporization of cannabis
  Other Names: marijuana

SUMMARY:
Acute cannabis administration is reported to alleviate HIV neuropathic pain (HIV-NP), but there is limited knowledge about the effects of cannabis constituents (delta-9 tetrahydrocannabinol/THC and cannabidiol/CBD), the consequences of long-term cannabis use, and the impact of cannabis on endocannabinoid (EC) function in people living with HIV- NP. Our objective is to address these three fundamental gaps in our knowledge by: 1) examining the acute effects of various CBD/THC products on HIV-NP, 2) utilizing a mHealth text messaging protocol, Individual Monitoring of Pain and Cannabis Taken (IMPACT) to monitor daily real-world cannabis use and changes in pain; and 3) studying the relationship between cannabinoids, EC biomarkers, and chronic neuropathic pain

DETAILED DESCRIPTION:
Our objective is to assess 120 community-dwelling people living with HIV who have neuropathic pain and are currently using cannabis. These participants will be enrolled in a study that consists of two phases:

Phase 1) This will involve a cross over study involving three different doses of vaporized cannabis that contain THC and varying concentrations of CBD:

* Low CBD session: 8 puffs of 1.9% THC + 0.01% CBD
* Medium CBD sessions: 4 puffs of 1.4% THC + 0.01% CBD plus 4 puffs of 1.4% THC + 5.1% CBD
* High CBD sessions: 8 puffs of 1.4% THC + 5.1% CBD

This phase will examine the acute effects of cannabis on pain intensity, blood endocannabinoid levels, and the relationship of pain with heart rate variability (HRV).

Phase 2) This phase will involve the association between dispensary-obtained cannabis and changes in pain reported via IMPACT, a mHealth text messaging program that will serve as a useful tool to monitor the relationship between pain and cannabis use. Text messaging is an effective method to modify health behaviors, monitor substance use, and track pain. Our group has recently demonstrated the feasibility of using short message service (SMS) texting to promote anti-retroviral therapy adherence and monitor daily methamphetamine (METH) use in persons living with HIV neuropathy with bipolar disorder or METH dependence.

ELIGIBILITY:
Inclusion Criteria:

1. the ability to provide informed consent
2. age 18 or older
3. HIV infection documented at the HNRP or assessed by an HIV test at screening;
4. a diagnosis of HIV sensory neuropathy
5. current use of cannabis
6. the ability to describe the THC and CBD content in the products they use, i.e., obtaining cannabis from dispensaries that list THC and CBD content
7. ability to respond to daily text message

Exclusion Criteria:

1. meeting criteria for current substance or alcohol dependence
2. traumatic brain injury
3. dementia or Alzheimer's disease
4. psychosis
5. a respiratory condition, i.e., pulmonary disease, that would be exacerbated by inhaling vaporized cannabis
6. history of cardiovascular disease, including myocardial infarction or stroke;
7. uncontrolled hypertension, defined as a systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure greater than 100 mm Hg
8. pregnancy, breastfeeding, or unwillingness to prevent pregnancy during the cannabis administration portion of the study (using birth control in female participants of child- bearing age)
9. unwillingness or inability to receive or respond to text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brook L Henry, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC Center for Medicinal Cannabis Research, UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator, Brook Henry PhD (blhenry@ucsd.edu), will supply individual participant data to other researchers after the project is completed.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabis Administration Sessions: Participants attend three daily sessions, separated by 3- to 5-day intervals, where they inhale cannabis products. At one session (Low CBD) they inhale 8 puffs of vaporized cannabis containing 1.9% THC + 0.01 CBD. At one session (Medium CBD) they inhale 8 puffs of vaporized cannabis where 4 puffs contain 1.9% THC + 0.01 CBD and 4 puffs will contain 1.4% THC + 5.1% CBD. At one session (High CBD) they inhale 8 puffs of vaporized cannabis containing 1.4% THC + 5.1% CBD. The order of the Low CBD, Medium CBD, and High CBD sessions is randomized.
  Cannabis: vaporization of cannabis
Period: Overall Study
Arm/Group | Cannabis Administration Sessions
Started | 5
Low CBD Session | 5
Medium CBD Session | 5
High CBD Session | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cannabis Administration Sessions
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Numerical Pain Rating Scale (NPRS)
Description: This is a scale from 0 to 10 indicating the self-reported level of pain. 0 is the minimum score, indicating no pain. 10 is the maximum score indicating highest level of pain.
Time Frame: Pain is measured once before they receive study medication and then 2 minutes after drug treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
Number analyzed (Participants) | 5 | 5 | 5
units on a scale
  Before Drug Administration | 2.2 (0.7) | 2.6 (1) | 2.8 (0.8)
  After Cannabis Administration | 1.4 (0.6) | 1.2 (0.6) | 1.2 (0.4)

2. Secondary Outcome: Phase 1 - Patient Global Impression of Change (PGIC)
Description: This is a 7-point ordinal scale that asks the participant to rate improvement in their pain after drug administration compared to before drug administration. The scale range is 1 to 7. A score of 1 indicates the greatest improvement (reduction) in pain. A score of 7 indicates that pain is worse.
Time Frame: The PGIC was measured two minutes after drug administration.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Medium CBD Session: In the morning, participants will inhale 8 puffs of vaporized cannabis 4 puffs will contain 1.9% THC + 0.01 CBD and 4 puffs will contain 1.4% THC + 5.1% CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Cannabis: vaporization of cannabis
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 2.8 (0.6) | 2.6 (0.4) | 3.4 (0.7)

3. Secondary Outcome: Phase 1 - Von Frey Test
Description: This test measures sensitivity to pain causes by physical contact with the skin. The von Frey filament is applied to the dorsum of the more painful foot until bending is observed for 3 seconds. Pain is rated using a visual analog score (VAS). The scale is 0 to 100, where 0 indicates no pain and 100 indicates the worst pain.
Time Frame: The von Frey test was administered before drug administration and two minutes after drug administration.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Low CBD Session: In the morning, participants will inhale 8 puffs of vaporized cannabis containing 1.9% THC + 0.09 CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Cannabis: vaporization of cannabis
- High CBD Session: In the morning, participants will inhale 8 puffs of vaporized cannabis containing 1.4% THC + 5.4% CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Cannabis: vaporization of cannabis
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
Number analyzed (Participants) | 5 | 5 | 5
units on a scale
  Before Drug Administration | 28 (11.1) | 13.4 (9.4) | 14.5 (6.4)
  After Cannabis Administration | 7.4 (3.8) | 10.8 (5.7) | 8.8 (5.1)

4. Secondary Outcome: Phase 1 - Marijuana Subscale (M-scale) of the Addiction Research Center Inventory (ARCI)
Description: The M-scale has 12 true/false statements describing the subjective effects of marijuana on participants after they take the drug. Each question is scored as 0 or 1. The scale ranges from 0 (minimum score) to 12 (maximum score). A lower score indicates that the participant is experiencing fewer side effects of the drug. A higher score indicates that the participant is experiencing more side effects of the drug. Reported side effects on this scale include dry mouth, slower movements, shaking hands, and having a pleasant feeling.
Time Frame: The M-scale was administered 2 minutes after drug treatment.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Low CBD Session: In the morning, participants will inhale 8 puffs of vaporized cannabis containing 1.9% THC + 0.01 CBD. They will then undergo experimental testing as described below under Outcome Measures.
  Cannabis: vaporization of cannabis
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 1.4 (0.5) | 3.2 (0.6) | 1.8 (0.4)

5. Secondary Outcome: Phase 1 - Levels of the Endocannabinoid Biomarker Anandamide (AEA)
Description: Anandamide levels in plasma were quantified using liquid chromatography-tandem mass spectrometry (LC/MS).
Time Frame: AEA was quantified 60 minutes after drug administration.
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/ml)
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
Number analyzed (Participants) | 5 | 5 | 5
nanograms per milliliter (ng/ml) | 0.52 (0.08) | 0.53 (0.16) | 0.49 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 6 hours following each drug administration.
Arm/Group | Low CBD Session | Medium CBD Session | High CBD Session
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low CBD Session (N=5) | Medium CBD Session (N=5) | High CBD Session (N=5)
Drowsiness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Dry Mouth (General disorders) | 2 (2) | 2 (2) | 2 (2)
Cognitive Impairment (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03099005/Prot_SAP_000.pdf